CLINICAL TRIAL: NCT02766543
Title: Evaluation of the TULSA-PRO MRI-Guided Transurethral Ultrasound Prostate Ablation Device in Patients With Localized Prostate Cancer: a Prospective, Single-Arm, Pivotal Clinical Study
Brief Title: Pivotal Study of MRI-guided Transurethral Ultrasound Ablation in Patients With Localized Prostate Cancer
Acronym: TACT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Profound Medical Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCP-10100
Record Dates: First submitted 2016-05-05; First posted 2016-05-09 (Estimated); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; high intensity transurethral ultrasound ablation; MRI-guided; minimally invasive; real-time temperature feedback control; whole-gland; TULSA
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MRI-guided Transurethral Ultrasound Ablation Device (Experimental): Magnetic resonance imaging-guided transurethral ultrasound ablation of whole-gland prostate tissue.
  Interventions: Device: MRI-guided Transurethral Ultrasound Ablation

INTERVENTIONS:
Device: MRI-guided Transurethral Ultrasound Ablation — Magnetic resonance imaging-guided transurethral ultrasound ablation is a novel minimally-invasive procedure where the therapeutic endpoint is prostate ablation through thermal coagulation.
  Other Names: TULSA-PRO

SUMMARY:
A prospective, multi-center, single-arm study, planned in 150 patients. The primary objective of the study is to further evaluate the safety and efficacy of a magnetic resonance imaging (MRI)-guided transurethral ultrasound therapy system (TULSA-PRO) intended to ablate prostate tissue of patients with localized, organ-confined prostate cancer.

DETAILED DESCRIPTION:
Profound Medical Inc. has developed a novel technology called the MRI-guided transurethral ultrasound therapy system (TULSA-PRO). The technology is developed for patients with organ confined prostate cancer. The therapeutic endpoint of this technology is thermal coagulation of prostate tissue.

The treatment is conducted within a MRI suite, which enables real-time temperature images of the heated region to be acquired as the ultrasonic treatment is delivered. Using MRI thermometry during treatment, dynamic temperature feedback control over the intensity of the ultrasound beams and rotation of the Ultrasound Applicator can shape the pattern of thermal coagulation accurately and precisely in the prostate gland.

It provides advantages of a non-invasive procedure with short treatment times.

ELIGIBILITY:
Inclusion Criteria:

1. Male, age 45 to 80 years
2. Biopsy-confirmed adenocarcinoma of the prostate. Biopsy (minimum 10 cores) obtained ≥ 6 weeks and ≤ 6 months before treatment (or at the discretion of PI and approval by the Sponsor).
3. Clinical stage ≤ T2b

4.1 Gleason score ≤ 3 + 4 (Part I only)

4.2 Gleason score 3+4 (Part II only) *now recruiting

5. PSA ≤ 15 ng/ml

6. Eligible for MRI [Form GCP-10131]

7. Eligible for general anesthesia (ASA category ≤ 3)

8. Prostate volume ≤ 90 cc, on Baseline MRI

9. Prostate size ≤ 5.0 cm in sagittal length, and ≤ 6.0 cm in axial diameter, on Baseline MRI

10. Life expectancy ≥ 10 years

11. No calcifications in the planned ultrasound beam path, or at the discretion of the investigator with approval from the Sponsor.

Exclusion Criteria:

1. Evidence (including Baseline MRI and bone scan) of extracapsular extension, sphincter involvement, seminal vesicle invasion, lymph node invasion or metastases
2. Suspected tumour on Baseline MRI within 3 mm of the prostatic urethra, or in the prostate apex within 3 mm from the sphincter plane
3. Prior definitive treatment of prostate cancer
4. Prior transurethral resection of the prostate (TURP)
5. Use of 5-alpha reductase inhibitors (5-ARIs) or hormone therapy within 3 months prior to the baseline visit. Baseline PSA must be established after a minimum of 3 months following 5-ARIs discontinuation. Additionally, use of 5-ARIs is not permitted following treatment during the study follow-up period.
6. Prostate calcifications > 1 cm in largest diameter, on Baseline Ultrasound
7. Cysts > 1 cm in largest diameter, on Baseline MRI
8. Bleeding disorder (INR > ULN and PTT > ULN)
9. Abnormal coagulation and current anticoagulant therapy. Patients whose anticoagulation therapy can be temporarily reversed within 7 days prior to treatment are eligible. Platelet inhibitors (ie: ASA) and heparin are not exclusion criteria.
10. Acute unresolved Urinary Tract Infection (UTI)
11. Interest in future fertility
12. History of any other malignancy other than skin cancer, or low grade bladder cancer which has been completely resected, within the previous 2 years. Patients that have had curative treatment of a previous malignancy and no recurrence of that malignancy within the past 2 years will be allowed.
13. Patients with peripheral arterial disease with intermittent claudication or Leriches Syndrome
14. Patients with diabetes who have evidence of complications from their diabetes, such as end organ sequelae of diabetes or Hemoglobin A1c > 7%.
15. History of any major rectal or pelvic surgery or radiotherapy
16. History of ulcerative colitis or other chronic inflammatory conditions affecting rectum (includes rectal fistula, anal stenosis)
17. Documented clinical prostatitis requiring therapy within 6 months prior to Treatment
18. History of urethral and bladder outlet disorders, including urethral stricture disease, urethral diverticulae, bladder neck contracture, urethral fistulae, urethral stenting, urethral sling, urethroplasty or chronic indwelling urethral catheter
19. Patients with artificial urinary sphincter or any penile implant
20. Severe neurogenic bladder
21. Untreated bladder stones
22. History of acute urinary retention within the last 12 months
23. Active untreated gross hematuria for any cause
24. Post Void Residual (PVR) bladder volume > 250 mL
25. Obstructing median lobe enlarged out of proportion to the rest of the prostate and protruding significantly into the bladder, sometimes referred to as "ball valve" median lobe, determined on Baseline MRI
26. Any prostate related investigational therapy within 6 months of Visit 1
27. History of Parkinson's disease or multiple sclerosis
28. History of drug abuse
29. Known infectious disease including HIV positivity or AIDS-related illness, HBV and HCV
30. Current unilateral or bilateral hydronephrosis
31. Allergy or contraindications to administration of the GI anti-spasmodic drug:

    1. Patients in the USA: Glucagon
    2. Patients in Canada and Europe: Buscopan (Hyoscine)
32. Contraindications to administration of gadolinium-based MRI contrast agent (e.g. Magnevist), such as chronic, severe kidney disease, acute kidney injury, history of Sickle Cell Disease, history of anemia, or intolerance/allergy to the contrast agent
33. Other severe, acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-09-21 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Safety Endpoint - Incidence of treatment-emergent adverse events | 1 year
  Frequency and severity of all adverse events will be evaluated by attribution and reported in accordance with the Common Terminology Criteria for Adverse Events (CTCAE) standard published by the National Cancer Institute (NCI).
Efficacy Endpoint - Proportion of patients achieving a PSA nadir ≤ 25% of the pre-treatment baseline value. | 1 year
  Prostate ablation efficacy will be evaluated using the proportion of patients achieving a PSA nadir ≤ 25% of the pre-treatment baseline value.

SECONDARY OUTCOMES:
Erectile Dysfunction Endpoint | At each visit post treatment throughout the total study follow-up - (1 month, 3 months, 6 months, 1 year, 2 years, 3 years, 4 years and 5 years).
  Rate of erectile dysfunction, determined by the change from baseline of the proportion of patients with IIEF-5 < 17.
Erection Firmness Endpoint | At each visit post treatment throughout the total study follow-up - (1 month, 3 months, 6 months, 1 year, 2 years, 3 years, 4 years and 5 years).
  Rate of erection firmness sufficient for penetration, determined by the change from baseline of the proportion of patients with IIEF item 2 ≥ 2.
Urinary Incontinence Endpoint | At each visit post treatment throughout the total study follow-up - (1 month, 3 months, 6 months, 1 year, 2 years, 3 years, 4 years and 5 years).
  Rate of urinary incontinence, determined by the change from baseline of the proportion of patients with EPIC item 5 ≥ 1 (one or more pads per day).
PSA Nadir Endpoint | 1 year
  Proportion of patients achieving PSA nadir ≤ 0.5 ng/ml.
PSA Stability Endpoint | At each visit post treatment throughout the total study follow-up - (1 month, 3 months, 6 months, 1 year, 2 years, 3 years, 4 years and 5 years).
  Proportion of patients with PSA ≤ 0.5 ng/ml at the most recent follow-up visit.
Prostate Volume Endpoint | 1 year
  Prostate volume reduction, evaluated on MRI between the treatment day and 12-month follow-up visits.
Prostate Biopsy Endpoint | 1 year
  Proportion of patients with negative prostate biopsy at the 12-month follow-up visit, determined by transrectal ultrasound-guided 10-core biopsy.
IPSS Endpoint | At each visit post treatment throughout the total study follow-up - (1 month, 3 months, 6 months, 1 year, 2 years, 3 years, 4 years and 5 years).
  Change in International Prostate Symptom Score (IPSS), between the baseline and most recent follow-up visit.
IIEF Endpoint | At each visit post treatment throughout the total study follow-up - (1 month, 3 months, 6 months, 1 year, 2 years, 3 years, 4 years and 5 years).
  Change in the Erectile Function, Orgasmic Function, Sexual Desire, Intercourse Satisfaction and Overall Satisfaction domains of the International Index of Erectile Function (IIEF-15), between the baseline and most recent follow-up visit.
EPIC Endpoint | At each visit post treatment throughout the total study follow-up - (1 month, 3 months, 6 months, 1 year, 2 years, 3 years, 4 years and 5 years).
  Change in Urinary, Bowel, Sexual and Hormonal domains of the Expanded Prostate Cancer Index Composite (EPIC), between the baseline and most recent follow-up visit.
Targeting Accuracy Endpoint | During treatment
  Conformal prostate ablation, measured quantitatively between the target prostate volume and the target temperature isotherm on MRI thermometry acquired during the TULSA-PRO procedure, and described using three measures of targeting accuracy (Dice Similarity Coefficient; Over- and under-targeted volumes; Linear targeting in mm).
CE-MRI Endpoint | Immediately after treatment
  Conformal prostate ablation, assessed qualitatively by visualizing the peripheral region of enhancement surrounding the non-perfused volume (NPV) on contrast-enhanced (CE)-MRI acquired immediately after treatment.
mpMRI Endpoint | 1 year
  Characterize the effect of the TULSA-PRO ablation on diagnostic multi-parametric prostate MRI (mpMRI), determined using PI-RADS v2 performed at the Baseline and 12-month follow-up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Eggener, MD, Principal Investigator — University of Chicago
Locations (14):
- United States (8):
  - University of California Los Angeles, Los Angeles, California
  - Yale Cancer Centre, New Haven, Connecticut
  - University of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Johns Hopkins Medicine, Baltimore, Maryland
  - William Beaumont Hospital, Royal Oak, Michigan
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
- Canada (2):
  - London Health Sciences Centre, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
- Germany (2):
  - University Hospital of Cologne, Cologne
  - Universitätsklinikum Heidelberg (University of Heidelberg, Dept of Urology), Heidelberg
- Radboud University Medical Center, Nijmegen, Netherlands
- ResoFus Alomar (Hospital Universitari De Bellvitge), Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wright C, Makela P, Bigot A, Anttinen M, Bostrom PJ, Blanco Sequeiros R. Deep learning prediction of non-perfused volume without contrast agents during prostate ablation therapy. Biomed Eng Lett. 2022 Nov 8;13(1):31-40. doi: 10.1007/s13534-022-00250-y. eCollection 2023 Feb. PMID 36711157
- See also: FDA 510k Summary — https://www.accessdata.fda.gov/cdrh_docs/pdf19/K191200.pdf

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/43/NCT02766543/Prot_SAP_001.pdf